CLINICAL TRIAL: NCT03380338
Title: Lifestyle Intervention in Patients With Diabetes Type 2 and the Association With the Gut Microbiota
Brief Title: The Effect of Exercise on Gut Microbiota in Type 2 Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Erik Serne, Principal Investigator, Amsterdam UMC, location VUmc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Bootcamp2
Record Dates: First submitted 2017-12-08; First posted 2017-12-21 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Type 2 Diabetes Mellitus; Insulin Sensitivity/Resistance
Keywords: Gut microbiota
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise program (Experimental): Twice weekly exercise program, combined aerobic and strenght training
  Interventions: Behavioral: Combined aerobic and strength exercise

INTERVENTIONS:
Behavioral: Combined aerobic and strength exercise

SUMMARY:
To investigate whether targeted lifestyle intervention (exercise), induces a change in intestinal fecal microbiota related to improved glycemic control and systemic inflammation in patients with DM type 2.

DETAILED DESCRIPTION:
Diet and exercise are the most beneficial lifestyle interventions in patients with diabetes mellitus (DM) type 2, causing an increase in glucose tolerance.

One of the mechanisms through which these treatment modalities work might be explained through changes in the gut microbiota. Recent studies show that the chronic inflammatory status causing insulin resistance in DM type 2, is triggered by an increase in circulating bacterial lipopolysaccharide (LPS). Strict lifestyle intervention, such as exercise, so called Diabetes Bootcamp (DB), may manipulate the gut microbiota, reducing circulating LPS, causing an improvement of the insulin-mediated

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet the criteria for diabetes type 2 (a random blood sugar of > 11.1 mmol/L and/or a fasting blood sugar lever of >7.0 mmol/L and/or a blood sugar of >11.1 mmol/L two hours after an oral glucose tolerance test and/or an HbA1c level of >47 mmol/mol).
* Male or female (post-menopausal)
* Age above 45 years and below 70 years
* BMI >30 kg/m2
* HbA1c < 80 mmol/mol or < 8,6% Subjects must use metformin
* Stable medication use
* Stable tension regulation (with or without medication)
* Subjects should be able to give informed consent

Exclusion Criteria:

* A history of cardiovascular event (Cerebrovascular event, myocardial infarction or pacemaker implantation)
* Severe-very severe lung emphysema (GOLD stage III-IV)
* Use of any antibiotics or proton pump inhibitor (PPI) in the past three months
* Use of any other antidiabetic medication besides metformin (e.g. SU-derivates, insulin)
* Use of a platelet inhibitor or cumarin derivate during
* Subjects participated in a lifestyle programme in the past 6 months (diet or exercise)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-05-11 (Actual); Primary Completion 2017-06-29 (Actual); Study Completion 2017-06-29 (Actual)

PRIMARY OUTCOMES:
Changes in gut microbiota composition upon exercise | At baseline, after 7 weeks, after 13 weeks
  alfa-diversity, beta-diversity
Change in insulin senistivity | Before and after exercise, i.e. from first visit (0 weeks) untill last visit (13 weeks)
  Rate of disappearance measured by the hyperinsulinemic-euglycemic clamp with stable glucose isotopes.
Change in capillary recruitment | Before and after exercise, i.e. from first visit (0 weeks) untill last visit (13 weeks)
  Insulin-induced capillary recruitment in skeletal muscle and heart

SECONDARY OUTCOMES:
Changes in resting energy expenditure | Before and after exercise
  Indirect calorimetry
Changes in continous cardiovascular monitoring | Before and after exercise

CONTACTS AND LOCATIONS:
Locations (1):
- VU University Medical Center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No